CLINICAL TRIAL: NCT04441086
Title: Emotion Regulation Intervention to Sustain Physical Activity in Rural-dwelling Women and Men After Myocardial Infarction
Acronym: eMotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other); Jonas Philanthropies (Unknown)
Responsible Party: Principal Investigator, Kelly L. Wierenga, Assistant Professor, Nursing, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2002325890
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Event; Emotions
Keywords: Emotion regulation
MeSH Terms: conditions — Cardiovascular Diseases; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: 3 group randomized control trial. Conditions include eMotion intervention, healthy living active control, and usual care.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eMotion (Experimental): The eMotion intervention is based on feasibility testing of the successful in-person program with critical refinement to improve accessibility. eMotion has undergone subsequent content validity testing with intervention development, self-management, cardiovascular health, and health information technology delivery experts. eMotion teaches a carefully selected repertoire of emotion regulation strategies well suited for aging rural adults following a first cardiac event in tandem with usual cardiac rehabilitation. The intervention helps patients recognize their emotions, balance emotional and physical wellbeing, and implement emotion regulation strategies effectively. Intervention provided in addition to usual cardiac rehabilitation.
  Interventions: Behavioral: eMotion
- Healthy living active control (Active Comparator): Healthy living strategies based on American Heart Association education. Intervention provided in addition to usual cardiac rehabilitation.
  Interventions: Behavioral: Healthy Living Active Control
- Usual care (No Intervention): Usual cardiac rehabilitation with no additional intervention.

INTERVENTIONS:
Behavioral: eMotion — Content is delivered within the context of emotion provoking situations common in those recovering from a first MI and in maintaining MVPA. The new on-demand access to asynchronous content sessions provides didactic presentation of video and written material based on weekly needs assessments. Weekly scheduled synchronous video chat sessions, led by a nurse interventionist, will provide further individualization and application of content materials.
  Arms: eMotion
Behavioral: Healthy Living Active Control — The attention control group will receive their usual cardiac rehabilitation and a comparable dose matched (to that of the eMotion intervention) of healthy living web content and video chat with a nurse.
  Arms: Healthy living active control

SUMMARY:
The purpose of this study is to evaluate early preliminary efficacy of the eMotion intervention in US adults who have experienced a first cardiac event and participating in phase II cardiac rehabilitation.

This study will evaluate early efficacy and evaluate the cognitive processes as intervention response variables. Investigators will also examine the relationships between emotion regulation and other cognitive processes and symptoms (threat and stress, cognition and motivation), symptoms [depression, anxiety, pain, sleep, and fatigue]), and health related quality of life among adults enrolled in cardiac rehabilitation after a first cardiac event.

DETAILED DESCRIPTION:
Aim 1: Evaluate early preliminary efficacy of the eMotion intervention

Research hypothesis 1. Compared with adults randomized to active healthy living attention control and usual care control groups, adults randomized to eMotion will have greater improvement in these outcomes over time:

1.1. Improved minutes of moderate to vigorous physical activity 1.2. Symptom improvement (depression, anxiety, pain, sleep, and fatigue) 1.3. Health related quality of life.

Aim 2: Evaluate the cognitive processes as intervention response variables.

Research hypothesis 2. Compared with adults randomized to active healthy living attention control and usual care control groups, adults randomized to eMotion will have:

2.1. Improved emotion regulation (efficiency and strategy use) 2.2. Decreased perceived cardiac threat and general stress 2.3. Improved cognition and motivation

Aim 3. Exploratory. Examine the relationships between emotion regulation and other cognitive processes and symptoms (threat and stress, cognition and motivation), and symptoms [depression, anxiety, pain, sleep, and fatigue]) among adults enrolled in cardiac rehabilitation after a first major cardiac event.

ELIGIBILITY:
Inclusion Criteria:

1. First time major cardiac event as documented in medical record;
2. enrolled in cardiac rehabilitation phase II program;
3. living independently; and
4. at least mild symptoms of depression and/or anxiety (determined by standardized measure cutpoints).

Exclusion criteria:

1. does not speak English;
2. major Axis 1 psychiatric diagnosis (e.g. schizophrenia);
3. terminal cancer; and
4. legally blind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Change in Moderate to Vigorous Physical Activity (MVPA) | 1 week trials at baseline, 12 weeks, 20 weeks, and 52 weeks
  Minutes spent in MVPA

SECONDARY OUTCOMES:
Change in Depression Symptoms | Baseline to 12 weeks, 20 weeks, and 52 weeks
  Symptoms of depression measured using the Depression, Anxiety, and Stress Scale (DASS)
Change in Anxiety Symptoms | Baseline to 12 weeks, 20 weeks, and 52 weeks
  Symptoms of anxiety measured using the Depression, Anxiety, and Stress Scale (DASS)
Change in Pain Symptoms | Baseline to 12 weeks, 20 weeks, and 52 weeks
  Pain will be measured with the Brief Pain Inventory
Change in Sleep efficiency | Baseline to 12 weeks, 20 weeks, and 52 weeks
  Sleep efficiency will be a calculation of the ratio of the total sleep time to time spent in bed using the ActiGraph wGT3X-BT accelerometer
Change in Fatigue Symptoms | Baseline to 12 weeks, 20 weeks, and 52 weeks
  Fatigue will be measured using the Fatigue Severity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L Wierenga, PhD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Indiana University Health West Hospital, Avon, Indiana
  - Indiana University Health Bedford Hospital, Bedford, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Health Tipton Hospital, Tipton, Indiana

REFERENCES:
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536